CLINICAL TRIAL: NCT04776720
Title: Ancillary Study of a Randomized Controlled Trial of a Group Based Therapeutic Yoga Intervention for Urinary Incontinence in Ambulatory Older Women
Brief Title: Ancillary Study of the Lessening Incontinence With Low-impact Activity Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K24AG068601 (NIH); 1R01DK116712-01A1 (NIH); K24AG068601 (NIH)
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Program (Experimental): The 3-month yoga intervention provides instruction and practice in a variety of yoga postures and techniques that have been selected by the study yoga expert consultants for their potential to improve bladder control and safety and feasibility for the target population.
  Interventions: Behavioral: Yoga Practice Program
- Physical Conditioning Program (Active Comparator): The 3-month physical conditioning program provides instruction and practice in a variety of exercises and stretches that have been designed by the study physical therapist.
  Interventions: Behavioral: Physical Conditioning Program

INTERVENTIONS:
Behavioral: Yoga Practice Program — 3 month group yoga classes
  Arms: Yoga Program
Behavioral: Physical Conditioning Program — 3 month group physical conditioning classes
  Arms: Physical Conditioning Program

SUMMARY:
The parent trial that supports this ancillary research is a randomized controlled trial to evaluate the efficacy of a group-based yoga intervention to decrease the frequency and impact of urinary incontinence in ambulatory middle-aged and older women.

Women aged 45 years and older who report daily or more frequent stress-, urgency-, or mixed-type incontinence, are not already engaged in formal yoga or muscle stretching/strengthening programs, are willing to temporarily forgo other clinical treatments for incontinence, are able to walk to and use the bathroom without assistance, and meet other eligibility criteria are being recruited from multiple locations surrounding the San Francisco Bay area. Following a series of telephone- and then clinic-based screening assessments, including a voiding diary to confirm the frequency and clinical type of incontinence, eligible women are randomized in a 1:1 ratio to participate in either a 3-month yoga program (N~120) or a time-equivalent, non-specific muscle stretching and strengthening control program (N~120).

During the 3-month intervention period, participants participate in structured intervention programs (either yoga-specific or muscle stretching-strengthening) consisting of twice weekly, 90-minute group classes led by trained instructors). They are also be instructed to practice their assigned intervention for at least an additional hour per week, with the assistance of participant manuals created by the study team and a set of home yoga or stretching/strengthening exercise props.

For this ancillary trial research, the investigators are examining ancillary measures of a) physical performance status, b)perceived stress, depression, and anxiety symptoms, and c) sleep quality, duration, and continuity, already incorporated by the principal investigator into the parent trial. The investigators will examine prospective relationships between these ancillary measures and participant-reported urinary incontinence frequency/severity/impact, examine intervention effects on these ancillary outcomes, and assess the extent to which these ancillary outcomes mediate intervention effects on incontinence frequency/severity/impact.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 45 years or older who report urinary incontinence starting at least 3 months prior to screening
* Self-report an average of at least one incontinence episodes per day voiding diary
* Self-report urgency-predominant (i.e., at least half of incontinence episodes being urgency-type), stress-predominant (i.e., at least half of episodes being stress-type), or mixed-type (i.e., an equal number of stress- and urgency-type episodes) incontinence on the screening voiding diary
* Willing to refrain from initiating medical treatments that may affect their incontinence or voiding pattern during the study intervention period

Exclusion Criteria:

* Current participation in organized yoga classes or workshops, or any prior organized yoga training directed specifically at improving incontinence
* Current participation in organized physical conditioning classes involving muscle strengthening exercises (e.g., Pilates)
* Current urinary tract infection or hematuria detected by urinalysis at screening visit (women can re-present after evaluation and treatment through their usual care)
* Report use of medical devices (i.e. pessary) for incontinence within the past month (participants may stop use of device and re-present for study)
* Report use of bladder botox, electrostimulation, formal bladder training, or formal pelvic floor exercise training (with certified practitioners) in the past 3 months
* Report any history of prior anti-incontinence or urethral surgery (not including urethral dilation), pelvic cancer, or pelvic irradiation
* Report other surgery to the pelvis (hysterectomy, oophorectomy, vaginal surgery, bladder surgery, colon surgery) within the past 3 months
* Unable to walk 2 blocks on level ground without assistance (functional capacity < 4 metabolic equivalents)
* Unable to get up from a supine to a standing position without assistance (assessed during the screening visit)
* Report history of interstitial cystitis, bladder or rectal fistula, or congenital defect causing urinary incontinence
* Report incontinence caused by a major neurologic conditions such as multiple sclerosis, spinal cord injury, or Parkinson's disease
* Report use of medications with strong effects on urination (anticholinergic bladder medications, beta-3 agonists, tricyclic antidepressants, mirabegron, loop diuretics) within the past month
* Report starting, stopping, or changing the dose of a medication with the potential to affect anxiety or depression symptoms (i.e., selective serotonin reuptake inhibitors, anxiolytics/sedatives, antipsychotics) within the past 1 month, or plans to start, stop, or change to dose of such a medication during the study period
* Participation in another research study that involves investigational drugs or devices that could potentially confound the results of this study
* Unable to understand study procedures, complete study interviews, or and provide informed consent in English
* Report conditions that, in the judgment of the investigators, render potential participants unlikely to follow the protocol, including plans to move, substance abuse, significant psychiatric problems, or dementia

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Huang, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hough E, Goldstein LA, Subak LL, Chesney MA, Schembri M, Raghunathan H, Balys Pawlowsky S, Huang AJ. Effects of Hatha Yoga vs Physical Conditioning on Sleep in Women With Urinary Incontinence: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2546499. doi: 10.1001/jamanetworkopen.2025.46499. PMID 41359336

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Yoga Program | Physical Conditioning Program
Started | 121 | 119
Completed | 101 | 109
Not Completed | 20 | 10
Not completed — COVID Related | 4 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Serious Adverse Event | 0 | 1
Not completed — Too Busy | 3 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Family | 2 | 2
Not completed — No remote technology access | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Cannot tolerate intervention | 1 | 0
Not completed — Incomplete outcome data | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yoga Program | Physical Conditioning Program | Total
Number analyzed (Participants) | 121 | 119 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.7) | 61.4 (8.8) | 62.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 119 | 240
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 83 | 77 | 160
  Black | 7 | 12 | 19
  Hispanic | 21 | 11 | 32
  Asian | 20 | 20 | 40
  Native Hawaiian or PI | 0 | 0 | 0
  American Indian | 0 | 0 | 0
  More than one race | 11 | 9 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 121 | 119 | 240
Total Urinary Incontinence Episodes [Mean (Standard Deviation); unit: episodes per day] | 3.6 (2.5) | 3.2 (1.9) | 3.4 (2.2)
Stress-Type Urinary Incontinence Episodes [Mean (Standard Deviation); unit: episodes per day] | 1.4 (1.8) | 1.4 (1.5) | 1.4 (1.6)
Urgency-Type Urinary Incontinence Episodes [Mean (Standard Deviation); unit: episodes per day] | 2.1 (2.2) | 1.7 (1.4) | 1.9 (1.9)
Incontinence Impact Questionnaire (IIQ) [Mean (Standard Deviation); unit: units on a scale] — Range 0-400, Higher score indicates lower quality of life
  units on a scale | 100.4 (78.9) | 101.6 (66.4) | 101.0 (72.7)
Urogenital distress inventory-6 score (UDI) [Mean (Standard Deviation); unit: units on a scale] — Range 0-100, Higher score indicates lower quality of life
  units on a scale | 39.1 (19.1) | 28.5 (19.4) | 38.8 (19.2)
Patient Perception of BladderCondition (PPBC) [Mean (Standard Deviation); unit: units on a scale] — Range 1-6, Higher score indicates lower quality of life
  units on a scale | 3.3 (1.0) | 3.4 (1.0) | 3.4 (1.0)
Center for Epidemiologic Studies Depression Scale (CES-D) [Mean (Standard Deviation); unit: units on a scale] — Range 0-60, Higher score indicates lower quality of life
  units on a scale | 10.1 (8.8) | 10.0 (8.1) | 10.0 (8.4)
State/Trait Anxiety Inventory (STAI)--Trait [Mean (Standard Deviation); unit: units on a scale] — Range 20-80, Higher score indicates lower quality of life
  units on a scale | 36.1 (11.2) | 36.1 (10.5) | 36.1 (10.9)
Hospital Anxiety & Depression (HADS)--Anxiety score [Mean (Standard Deviation); unit: units on a scale] — Range 0-21, Higher score indicates lower quality of life
  units on a scale | 5.3 (3.8) | 5.2 (3.7) | 5.3 (3.8)
Perceived Stress Scale (PSS) score [Mean (Standard Deviation); unit: units on a scale] — Range 0-40, Higher score indicates lower quality of life
  units on a scale | 13.0 (7.2) | 13.3 (6.8) | 13.2 (7.0)
PROMIS Physical 8B, T-Score [Mean (Standard Deviation); unit: T-score] — (mean 50, Std Dev 10) no widely accepted thresholds have been published Higher score indicates better quality of life
  T-score | 51.0 (6.2) | 51.3 (6.8) | 51.2 (6.5)
One-legged Balance Test [Mean (Standard Deviation); unit: seconds] — Range 0-30, Higher score indicates better quality of life
  seconds | 24.4 (9.9) | 25.5 (8.7) | 24.9 (9.4)
Chair Stands (in 30 seconds) [Mean (Standard Deviation); unit: chair stands] — Higher score indicates better quality of life
  chair stands | 12.6 (3.9) | 13.1 (4.2) | 12.9 (4.1)
2-Minute Step Test [Mean (Standard Deviation); unit: steps] — Higher score indicates better quality of life
  steps | 85.9 (22.8) | 88.5 (26.1) | 87.2 (24.5)
Wake after sleep onset [Mean (Standard Deviation); unit: Minutes] — Higher score indicates lower quality of life
  Minutes | 24.4 (29.2) | 25.2 (25.6) | 24.8 (27.4)
Total sleep time [Mean (Standard Deviation); unit: hours] — Higher score indicates better quality of life
  hours | 7.1 (1.2) | 7.0 (1.0) | 7.0 (1.1)
Pittsburgh Sleep Quality Index (PSQI) total score [Mean (Standard Deviation); unit: units on a scale] — Range 0-21, Higher score indicates lower quality of life
  units on a scale | 6.2 (3.1) | 6.6 (3.1) | 6.4 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in One-legged Balance Test (Winsorized)
Description: Assess change in successive semi-tandem, tandem, and one-legged balance stand tests, in which their ability to hold each position for up to 30 seconds. Scoring is based on the number of seconds in which the participant is able to hold the one-legged balance position, ranging from 0 to 30. If a participant cannot make it through the semi-tandem and tandem stands, the one-legged balance will not be attempted. They will receive a score of zero for the one-legged balance.
  Change was calculated as the followup value minus the baseline value. Change values were Winsorized at the 1st and 99th percentile. Values are model generated Least Square Means for combined 6 and 12 week time points
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 107 | 110
seconds | 1.34 [0.52 to 2.16] | 1.53 [0.72 to 2.35]
Statistical Analysis 1: Comparison: Yoga Program vs Physical Conditioning Program; Test type: Superiority; p = 0.743, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 0.19, 95% CI 2-sided [-0.95 to 1.34]

2. Primary Outcome: Change From Baseline in Chair Stands (in 30 Seconds)
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points.
  Higher score indicates better quality of life
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: chair stands
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 105 | 106
chair stands | 1 [0.32 to 1.68] | 1.98 [1.3 to 2.66]
Statistical Analysis 1: Comparison: Yoga Program vs Physical Conditioning Program; Test type: Superiority; p = 0.043, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 0.98, 95% CI 2-sided [0.03 to 1.93]

3. Primary Outcome: Change From Baseline in 2-Minute Step Test
Description: Assess change in aerobic endurance. In this test of aerobic endurance for older adults, participants are asked to step in place as many times as possible in a 2 minute period, each time raising the knee to a level midway between the patella and iliac crest.
  Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points Higher scores indicating greater endurance.
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: steps
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 104 | 109
steps | 8.05 [4.58 to 11.51] | 9.03 [5.59 to 12.48]
Statistical Analysis 1: Comparison: Yoga Program vs Physical Conditioning Program; Test type: Superiority; p = 0.689, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, with variance co-variance matrix; Model based LS mean difference = 0.99, 95% CI 2-sided [-3.87 to 5.84]

4. Secondary Outcome: Change From Baseline in Perceived Stress Scale (PSS) Score
Description: Assess change in total score on Perceived Stress Scale (PSS), a 10-item measure of thoughts and feelings related to perceived stress in the past month, validated in a probability sample of the United States. Scores range from 0 to 40; higher scores indicated greater perceived stress.
  Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 106 | 112
units on a scale | -0.44 [-1.41 to 0.52] | -0.72 [-1.68 to 0.24]
Statistical Analysis 1: Comparison: Yoga Program vs Physical Conditioning Program; Test type: Superiority; p = 0.685, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -0.28, 95% CI 2-sided [-1.63 to 1.07]

5. Secondary Outcome: Change From Baseline in Center for Epidemiologic Studies Depression Scale (CES-D)
Description: Assess change in total score on Center for Epidemiologic Studies Depression (CES-D) scale, a validated 20-item self-administered questionnaire measure that has been widely used in clinical trials, including trials of bladder interventions, and has been shown to be sensitive to change. Total scores range from 0 to 60, with higher scores indicate greater burden of depression symptoms.
  Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 107 | 112
units on a scale | -0.82 [-2.25 to 0.6] | -0.52 [-1.93 to 0.9]
Statistical Analysis 1: Comparison: Yoga Program vs Physical Conditioning Program; Test type: Superiority; p = 0.764, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 0.3, 95% CI 2-sided [-1.69 to 2.3]

6. Secondary Outcome: Change From Baseline in State/Trait Anxiety Inventory (STAI)--Trait
Description: Assess change in somatic anxiety. Somatic anxiety (i.e., the affective component of anxiety believed to be related to autonomic physiological arousal response) is measured using the trait component of the Spielberger State Trait Anxiety Inventory (STAI), a 20-item self-administered measure validated in clinical populations, including patients with bladder symptoms. Scores range from 20 to 80, with higher scores indicating greater somatic anxiety.
  Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 107 | 112
score on a scale | -1.22 [-2.41 to -0.03] | -1.34 [-2.52 to -0.17]
Statistical Analysis 1: Comparison: Yoga Program vs Physical Conditioning Program; Test type: Superiority; p = 0.883, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -0.12, 95% CI 2-sided [-1.78 to 1.53]

7. Secondary Outcome: Change From Baseline in Hospital Anxiety & Depression (HADS)--Anxiety Score
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points. Range 0-21, Higher score indicates lower quality of life
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 107 | 111
units on a scale | -0.21 [-0.72 to 0.3] | -0.33 [-0.83 to 0.18]
Statistical Analysis 1: Comparison: Yoga Program vs Physical Conditioning Program; Test type: Superiority; p = 0.753, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -0.11, 95% CI 2-sided [-0.83 to 0.6]

8. Secondary Outcome: Change From Baseline in Wake After Sleep Onset (Winsorized)
Description: Assess change in sleep disruption. Average time spent awake after initial sleep onset is also assessed using the Pittsburgh Sleep Diary, based on participant recordings of nocturnal awakenings after initially falling asleep.
  Change was calculated as the followup value minus the baseline value. Change values were Winsorized at the 1st and 99th percentile. Values are model generated Least Square Means for combined 6 and 12 week time points. Higher score indicates lower quality of life.
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 104 | 108
minutes | -3.55 [-7.96 to 0.85] | -6.96 [-11.3 to -2.61]
Statistical Analysis 1: Comparison: Yoga Program vs Physical Conditioning Program; Test type: Superiority; p = 0.276, Mixed Models Analysis; Adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -3.4, 95% CI 2-sided [-9.54 to 2.74]

9. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) Total Score
Description: Assess change in global sleep quality. Subjective sleep quality is being assessed using the Pittsburgh Sleep Quality Index (PSQI), an 18-item validated questionnaire originally designed to assess sleep quality, latency, efficiency, and problems over a one-week period. A global sleep quality score ranging from 0 to 21 can be derived from the PSQI, with higher scores reflecting poor sleep quality.
  Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 108 | 112
units on a scale | -0.37 [-0.78 to 0.04] | -0.66 [-1.07 to -0.25]
Statistical Analysis 1: Comparison: Yoga Program vs Physical Conditioning Program; Test type: Superiority; p = 0.319, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -0.29, 95% CI 2-sided [-0.86 to 0.28]

10. Secondary Outcome: Change From Baseline in Total Sleep Time
Description: Assess change in average nightly sleep duration. Average total sleep duration is assessed using the Pittsburgh Sleep Diary is a daily self-report measure previously validated against actigraphy data, and used in multiple past studies of older adults.
  Change from baseline in Total sleep time. Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points.
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: hours
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 104 | 109
hours | 0 [-0.18 to 0.17] | 0.09 [-0.08 to 0.27]
Statistical Analysis 1: Comparison: Yoga Program vs Physical Conditioning Program; Test type: Superiority; p = 0.448, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 0.1, 95% CI 2-sided [-0.15 to 0.34]

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Yoga Program | Physical Conditioning Program
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/119
Serious Adverse Events (participants affected / at risk) | 1/121 | 1/119
Other Adverse Events (participants affected / at risk) | 37/121 | 43/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga Program (N=121) | Physical Conditioning Program (N=119)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
High Grade B-Cell Lymphoma Burkitt-Like Lymphoma Nos (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga Program (N=121) | Physical Conditioning Program (N=119)
Recurrent Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Detached Retina (Eye disorders) | 0 (0) | 1 (1)
Abdominal Cramps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 2 (2) | 2 (2)
Tooth Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Facial Pain (General disorders) | 0 (0) | 1 (1)
Allergy (Immune system disorders) | 1 (1) | 0 (0)
Allergy Nos (Immune system disorders) | 0 (0) | 1 (1)
Hay Fever (Immune system disorders) | 1 (1) | 0 (0)
Bladder Infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Coronavirus Infection (Infections and infestations) | 1 (1) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0)
Lower Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Mumps (Infections and infestations) | 1 (1) | 0 (0)
Shingles (Infections and infestations) | 1 (1) | 1 (1)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 4 (4) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Back Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Knee Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lateral Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Leg Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulled Hamstring (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shoulder Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toe Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaccination Adverse Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Colonoscopy (Investigations) | 1 (1) | 0 (0)
Endoscopy (Investigations) | 0 (0) | 1 (1)
Back Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Back Pain; Knee Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Frozen Shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hand Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hip Arthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hip Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Knee Swelling (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Leg Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Lumbar Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain Ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Elbow (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Patellofemoral Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator Cuff Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shoulder Deformity Nos (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Shoulder Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal Disorder Nos (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervical Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Localised Numbness (Nervous system disorders) | 1 (1) | 0 (0)
Migraine, Unspecified (Nervous system disorders) | 1 (1) | 0 (0)
Neck Numbness (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica Aggravated (Nervous system disorders) | 1 (1) | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma Aggravated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthmatic Attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cyst Epidermal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neck Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Back Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder Sling Procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Bunionectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee Arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Oral Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Shoulder Replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Hot Flashes (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT04776720/Prot_SAP_000.pdf